CLINICAL TRIAL: NCT04354831
Title: An Open Label, Phase 2 Study Evaluating the Efficacy and Safety of High-Titer Anti-SARS-CoV-2 Plasma in Hospitalized Patients With COVID-19 Infection
Brief Title: Efficacy and Safety of Convalescent Plasma in Treating COVID-19 Hospitalized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Froedtert Hospital (Other)
Responsible Party: Principal Investigator, Mary Beth Graham, MD, Associate Chief, Professor Infectious Disease, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037712
Record Dates: First submitted 2020-04-14; First posted 2020-04-21 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 131 patients in 2 cohorts (ICU cohort and a hospitalized non-ICU cohort)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICU Cohort (Experimental): Patients who are in the ICU at the time of enrollment. Patients will receive anti-SARS-CoV-2 convalescent plasma.
  Interventions: Biological: anti-SARS-CoV-2 convalescent plasma
- Non-ICU Cohort (Experimental): Patients who are NOT in the ICU at the time of enrollment. Patients will receive anti-SARS-CoV-2 convalescent plasma.
  Interventions: Biological: anti-SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: anti-SARS-CoV-2 convalescent plasma — * SARS-CoV-2 convalescent plasma (1-2 units; ~200-400 mL maximum dose as 7 ml/kg adjusted IBW )
  * Study drug will be administered as a single intravenous infusion

SUMMARY:
This is a Phase II study. This research study is being conducted to use convalescent donor plasma in seriously ill patients who have COVID-19.

DETAILED DESCRIPTION:
This is an open label phase 2 trial assessing the efficacy and safety of anti-SARS-CoV-2 convalescent plasma in hospitalized patients with acute severe respiratory symptoms from COVID-19. Symptomatic patients with clinical or radiological interstitial COVID-19 pneumonia and within 21 days of onset of symptoms will be enrolled in 2 cohorts - an ICU cohort and a hospitalized non-ICU cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years or older
2. Hospitalized as an in-patient with positive COVID-19 test by PCR
3. Presence of respiratory symptoms with any of severe features as below:

   * Respiratory Rate ≥ 24/min
   * Oxygen Support >3L/min by nasal cannula
   * New onset or worsening of respiratory symptoms with radiologic confirmation of bilateral ground glass opacities that cannot be attributed to another cause
4. Patient / HCPOA must agree to storage of blood specimens for future testing.
5. Patient / HCPOA is willing and able to provide electronic informed consent and comply with all protocol requirements. If patient is unable to consent due to incapacity, health care POA should be defined and able to consent for the patient.
6. Patients are allowed to receive all standard of care. Co enrollment in other clinical trials is permitted.

Exclusion Criteria:

1. FCBP with positive pregnancy test (mandatory)
2. Breastfeeding females
3. Receipt of pooled immunoglobulin (e.g. IVIG or other hyperimmune globulin products) in past 14 days. This does not apply to monoclonal antibodies .
4. Mechanical ventilation for > 14 days
5. Days from symptom onset >21 days
6. Expected survival < 72 hours
7. Contraindication to transfusion or history of prior reactions to transfusion blood products including any proven history of TRALI
8. Patients who were previously admitted to ICU cannot be enrolled in the non-ICU cohort. These patients could need ICU level care subsequently and at that time point could be considered for ICU cohort .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Graham, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ICU Cohort: Patients who are in the ICU at the time of enrollment. Patients will receive anti-SARS-CoV-2 convalescent plasma.
  anti-SARS-CoV-2 convalescent plasma: • SARS-CoV-2 convalescent plasma (1-2 units; ~200-400 mL maximum dose as 7 ml/kg adjusted IBW )
  • Study drug will be administered as a single intravenous infusion
- Non-ICU Cohort: Patients who are NOT in the ICU at the time of enrollment. Patients will receive anti-SARS-CoV-2 convalescent plasma.
  anti-SARS-CoV-2 convalescent plasma: • SARS-CoV-2 convalescent plasma (1-2 units; ~200-400 mL maximum dose as 7 ml/kg adjusted IBW )
  • Study drug will be administered as a single intravenous infusion
Period: Overall Study
Arm/Group | ICU Cohort | Non-ICU Cohort
Started | 41 | 90
Completed | 41 | 89
Not Completed | 0 | 1
Not completed — No blood type specific convalescent plasma was available | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICU Cohort | Non-ICU Cohort | Total
Number analyzed (Participants) | 41 | 90 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 60 | 89
  >=65 years | 12 | 30 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 43 | 64
  Male | 20 | 47 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 36 | 85 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 7 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 26 | 40
  White | 21 | 54 | 75
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 41 | 90 | 131
BMI [Mean (Full Range); unit: kg/m^2] | 35.34 [21.99 to 67.29] | 34.49 [18 to 64.64] | 34.76 [18 to 67.29]

OUTCOME MEASURES:

1. Primary Outcome: Overall Mortality
Description: Overall mortality during hospitalization for COVID-19. All patients were followed for the duration of their hospitalization, sometimes exceeding 60 days, through study completion.
Time Frame: Duration of patient hospitalization, sometimes exceeding 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | ICU Cohort | Non-ICU Cohort
Number analyzed (Participants) | 41 | 89
Participants | 22 | 7

2. Secondary Outcome: Length of Admission After Plasma Infusion
Description: Length of admission after convalescent plasma infusion for all patients. All enrolled patients, whether they were in the ICU cohort or in the non-ICU cohort, were monitored from the time of consent until the time of hospital discharge. Hospital discharge includes those patients who left the hospital alive and those patients who died during their stay.
Time Frame: Length of admission for COVID through study follow-up period
Measure: Mean (Full Range); unit: days
Arm/Group | ICU Cohort | Non-ICU Cohort
Number analyzed (Participants) | 41 | 89
days | 13.24 [1 to 66] | 7.85 [1 to 76]

3. Secondary Outcome: Length of ICU Stay After Convalescent Plasma Infusion
Description: Length of ICU stay after plasma infusion for patients who were in the experimental ICU cohort
Time Frame: Length of admission in the ICU for COVID through study follow-up period
Population: Only patients in the ICU Cohort were assessed for this outcome measure
Measure: Mean (Full Range); unit: days
Arm/Group | ICU Cohort
Number analyzed (Participants) | 41
days | 11.98 [1 to 66]

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events from the time of plasma infusion through the duration of their hospitalization, sometimes exceeding 60 days, through study completion.
Arm/Group | ICU Cohort | Non-ICU Cohort
All-Cause Mortality (participants affected / at risk) | 21/41 | 7/89
Serious Adverse Events (participants affected / at risk) | 12/41 | 14/89
Other Adverse Events (participants affected / at risk) | 0/41 | 4/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICU Cohort (N=41) | Non-ICU Cohort (N=89)
Bacteremia (Infections and infestations) | 4 | 1 — Patients who developed bacteremia during the hospital stay after enrollment and plasma infusion (not directly related to plasma infusion)
ICU Transfer (Respiratory, thoracic and mediastinal disorders) | 0 | 14 — Patients requiring ICU transfer after enrollment and plasma infusion (not directly related to plasma infustion)
Intubation (Respiratory, thoracic and mediastinal disorders) | 11 | 7 — Required intubation after enrollment and plasma infusion during the hospital stay (not directly related to plasma infusion)
Dialysis (Renal and urinary disorders) | 0 | 1 — Developed renal failure after enrollment and plasma infusion during hospitalization requiring dialysis (not related to plasma infusion)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICU Cohort (N=41) | Non-ICU Cohort (N=89)
Fever (General disorders) | 0 (0) | 2 (2) — Fever developed during infusion of convalescent plasma
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Rash developed within 72 hours of plasma infusion

LIMITATIONS AND CAVEATS:
Limitations: The plan was to infuse high titer plasma. All units were screened for SARS-CoV-2 antibody and were positive, but our blood bank was not able to provide specific titer information for each unit. We planned to monitor patients for up to 60 days post infusion, but once discharged pandemic concerns prevented follow-up.

Caveats: Inpatients were followed for duration of hospitalization, sometimes exceeding 60 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04354831/Prot_SAP_000.pdf